CLINICAL TRIAL: NCT00896701
Title: A Study of the Relationship Between Natural Killer Cell Recognition and Lysis of Autologous Leukemic Blasts and Clinical Outcome of Acute Myeloid Leukemia Patients Treated With Interleukin-2: A CALGB Leukemia Tissue Bank Project
Brief Title: Relationship Between Natural Killer Cells' Ability to Kill Leukemia Cells and the Outcome of Patients With Acute Myeloid Leukemia Previously Treated With Interleukin-2
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20206; CDR0000352018 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Flow Cytometry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow blast cells peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient samples from C9621, C9720 and C19808: This is a CALGB Leukemia Tissue Bank project that makes use of tissue from patients who have previously provided their consent. Diagnostic and follow-up samples from acute myeloid leukemia (AML) patients treated on CALGB protocols 9621, 9720 and 19808, and who have been registered on the mandatory companion Leukemia Tissue Bank Protocol CALGB 9665 will be used.
  Interventions: Other: flow cytometry; Other: immunologic technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: flow cytometry
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors predict response in patients previously treated with interleukin-2.

PURPOSE: This laboratory study is looking at the relationship between natural killer cells' ability to kill leukemia cells and the outcome of patients with acute myeloid leukemia previously treated with interleukin-2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate the in vitro lysis of autologous pre-treatment leukemic blast cells by interleukin-2 (IL-2)-expanded natural killer (NK) cells with relapse-free survival of patients with acute myeloid leukemia (AML) who were treated with interleukin-2 (IL-2).
* Correlate the expression of inhibitory (MHC class I) and activating ligands on AML blast cells with relapse-free survival of these patients.
* Correlate the expression of activating and inhibitory NK receptors on IL-2-expanded cells with relapse-free survival of these patients.
* Compare the susceptibility to autologous NK cell lysis of leukemic blasts obtained at diagnosis with those blasts obtained at relapse of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 60 vs ≥ 60 years) and cytogenetic risk category (favorable vs average vs poor).

Previously banked tissue samples of leukemic blast cells from bone marrow and natural killer (NK) cells from peripheral blood mononuclear cells are thawed and analyzed. Surface expression on leukemic blasts of co-stimulatory molecules, known activating NKG2D ligands, and MHC class I inhibitory ligands to NK cell receptors are quantified by monoclonal antibody analysis and flow cytometry. Mean cell fluorescence intensity (MCFI) of each ligand is correlated with relapse-free survival of the patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Prior treatment with interleukin-2 required
* Previously enrolled on CLB-9621, CLB-9720, or CALGB-19808
* Previously consented to companion Leukemia Tissue Bank Protocol CALGB-9665 and stored the following specimens:

  * Bone marrow blast cells procured at diagnosis and at relapse (when available)
  * Peripheral blood mononuclear cells obtained in remission

PATIENT CHARACTERISTICS:

Age

* 15 and over

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a CALGB Leukemia Tissue Bank project that makes use of tissue from patients who have previously provided their consent. Diagnostic and follow-up samples from acute myeloid leukemia (AML) patients treated on CALGB protocols 9621, 9720 and 19808, and who have been registered on the mandatory companion Leukemia Tissue Bank Protocol CALGB 9665 will be used.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2004-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Correlation of in vitro lysis of autologous pre-treatment acute myeloid leukemia (AML) blasts with relapse-free survival | Up to 10 years
Correlation of expression of inhibitory and activating ligands on AML blast cells with relapse-free survival | Up to 10 years
Correlation of expression of activating and inhibitory natural killer (NK) receptors on interleukin-2-expanded cells with relapse-free survival | Up to 10 years
Comparison of the susceptibility to autologous NK cell lysis of leukemic blasts obtained at diagnosis with those blasts obtained at relapse | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S. Farag, MD, PhD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (2):
- United States (2):
  - Kinston Medical Specialists, Kinston, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio